CLINICAL TRIAL: NCT06044649
Title: Comparative Mechanisms (Moderators, Mediators) of Psychosocial Treatments of Chronic Pain
Brief Title: Moderators and Mediators (M & M Trial) of Psychosocial Treatments of Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22010705
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain; Neck Pain; Back Pain
MeSH Terms: conditions — Chronic Pain; Neck Pain; Back Pain | interventions — Cognitive Behavioral Therapy; Acceptance and Commitment Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: 4-arm parallel randomized clinical trial comparing three therapies with each other and with a treatment as usual control
Who Masked: Outcomes Assessor
Masking Description: Masking of research staff and participants until baseline assessment is completed. Masking of research staff who interact with patients for outcome assessments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive Behavioral Therapy (Experimental): 8-session, individual, Cognitive Behavioral Therapy delivered remotely by skilled CBT therapists
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Acceptance and Commitment Therapy (Experimental): 8-session, individual, Acceptance and Commitment Therapy delivered remotely by skilled ACT therapists
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Emotional Awareness and Expression Therapy (Experimental): 8-session, individual, Emotional Awareness and Expression Therapy delivered remotely by skilled EAET
  Interventions: Behavioral: Emotional Awareness and Expression Therapy
- Treatment As Usual (Other): In this control condition, participants will engage in their usual care for neck/back pain with no additional experimental intervention
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — CBT endorses a pain management model and teaches people skills to cope with chronic pain.
  Other Names: CBT for chronic pain
  Arms: Cognitive Behavioral Therapy
Behavioral: Acceptance and Commitment Therapy — ACT is based on an acceptance model that seeks to decrease pain avoidance behaviors and enhance engagement in valued, adaptive activities that contribute to fewer pain-related restrictions in functioning.
  Other Names: ACT for chronic pain
  Arms: Acceptance and Commitment Therapy
Behavioral: Emotional Awareness and Expression Therapy — EAET advocates a pain treatment model in which pain can be substantially reduced by helping people learn that their pain is brain-based and can be substantially reduced or eliminated by decreasing fear of pain and of various emotional/interpersonal problems.
  Other Names: EAET for chronic pain
  Arms: Emotional Awareness and Expression Therapy
Other: Treatment as Usual — Participants assigned to TAU will not receive any additional psychosocial treatment beyond the other treatments they were receiving before enrolling in this study.
  Other Names: TAU
  Arms: Treatment As Usual

SUMMARY:
Chronic musculoskeletal pain (CP) is a major public health concern. Psychosocial treatments have been shown to be efficacious when compared to largely inert control conditions, but they are characterized by modest effects on primary outcomes. One strategy to boost efficacy is to increase our understanding of treatment mediators. Studies of mediators that directly compare different treatments with each other are needed to determine which mediators are treatment-specific, which are shared across treatments, and which contribute the most to clinical outcomes. Another strategy is to identify the patient characteristics that moderate treatment responses. Research is needed that is guided by theoretical models and that tests moderators across multiple treatments. Identifying subgroups of patients more likely to respond to one or another treatment can advance precision medicine by informing a priori patient-treatment matches that can optimize treatment effects. To accomplish these goals, the authors will conduct a randomized clinical trial to compare the mediators and moderators of the clinical effects of Cognitive-Behavioral Therapy (CBT), Acceptance and Commitment Therapy (ACT), and Emotional Awareness and Expression Therapy (EAET) on adults with chronic spinal (axial) pain. Following baseline assessment of outcome variables as well as potential mediators and moderators, 460 participants will be randomized to CBT, ACT, EAET, or treatment-as-usual control (TAU). The three treatments will be conducted as individual therapy provided weekly for 8 weeks via telehealth. The researchers will conduct weekly assessments of both potential mediators and outcomes, as well as post-treatment and 6-month follow-up assessments. The goal of the study is to identify the most powerful treatment mechanisms - specific and shared -- and reveal for whom the mediator-outcome pathways are strongest.This project can increase the effects of our psychosocial chronic pain treatments by identifying the most effective treatment mechanisms and by informing patient-treatment matches that can optimize treatment effects.

DETAILED DESCRIPTION:
Chronic musculoskeletal pain (CP) is a major public health concern. A number of psychosocial treatments have emerged in recent decades to help address this problem. These interventions have been shown to be efficacious when compared to largely inert control conditions; however, recent meta-analyses indicate that most of these treatments are characterized by modest effects on primary outcomes. This is a critical shortcoming of these otherwise promising approaches. Rather than attempting to boost efficacy only by developing new and hopefully more powerful interventions, we can also look within our already proven treatments for ways to enhance the magnitude of treatment effects. One strategy is to increase our understanding of treatment mediators. Studies of mediators that directly compare different treatments with each other are needed to determine which mediators are treatment-specific, which are shared across treatments, and which contribute the most to clinical outcomes. The findings from such research could be used to inform adaptations to existing treatment that enhance their benefits. A second strategy for increasing the beneficial effects of existing treatments is to identify the patient characteristics that moderate treatment responses. Research is needed that is guided by theoretical models and that tests moderators across multiple treatments. Identifying subgroups of patients more likely to respond to one or another treatment can advance precision medicine by informing a priori patient-treatment matches that can optimize treatment effects. To accomplish these goals, we will conduct a randomized clinical trial to compare the mediators and moderators of the clinical effects of Cognitive-Behavioral Therapy (CBT), Acceptance and Commitment Therapy (ACT), and Emotional Awareness and Expression Therapy (EAET) on adults with chronic spinal (axial) pain. Following baseline assessment of outcome variables as well as potential mediators and moderators we will randomize 460 participants to CBT, ACT, EAET, or treatment-as-usual control (TAU). The three treatments will be conducted as individual therapy provided weekly for 8 weeks via telehealth. We will conduct weekly assessments of both potential mediators and outcomes, as well as post-treatment and 6-month follow-up assessments. In addition to comparing the three treatments to each other (and TAU) for overall efficacy, we focus on two specific aims: Aim 1 is to identify mediators that are specific to treatments and those that are shared across treatments. Aim 2 is to identify baseline moderators of specific treatments and general predictors across treatments. This project can increase the effects of our psychosocial chronic pain treatments by identifying the most powerful treatment mechanisms - specific and shared -- and revealing for whom the mediator-outcome pathways are strongest. Via increased understanding of mediator and moderators, more effective pain treatment approaches can be developed, tested, and implemented.

ELIGIBILITY:
Inclusion Criteria:

* Back/neck is primary pain location (e.g., back/neck pain greater than leg pain)
* Pain for at least 3 months and experienced 4 or more days/week for the past 6 months
* Pain intensity last week is >= 3 (0 to 10 rating scale)
* Pain interference last week is >= 3 (0 to 10 rating scale)
* At least age 18
* Lives in United States
* Fluent in English
* Has personal computer/tablet and internet access
* Able to attend weekly sessions
* Willing to be randomized
* Seeking to improve their pain-related status via a psychological therapy

Exclusion Criteria:

Past 2 years (treated for or having experienced):

* Complex regional pain syndrome
* Epilepsy/seizure disorder
* Autoimmune disease
* Liver disease
* Cancer
* Heart disease
* Substance dependence or use disorder
* Schizophrenia or other psychotic disorder
* Bipolar disorder
* Obsessive-compulsive disorder
* Borderline personality disorder
* Suicide attempt or suicide intention or impulse

Also:

* Major medical procedure scheduled within next 9 months
* Applied for/ litigating for pain-related disability/worker's compensation (past year).
* Major life event/stressor in past 6 months
* Cognitive impairment (screener score <=4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) - Pain Severity | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  4-item measure of pain severity over past week (range 0 to 10; higher scores = worse pain severity)
Patient-Reported Outcome Measurement Information System (PROMIS) - Pain Interference - Short Form 8a | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  8-item measure of pain interference over past week (range1 to 5; higher scores = more pain interference)

SECONDARY OUTCOMES:
Patient Global Impression of Change | Weekly during treatment to post-treatment and 6-month follow-up
  1-item measure of overall health change since the start of the study (range 1 to 7; higher scores = more health improvement)
Patient-Reported Outcome Measurement Information System (PROMIS) - Physical Function - Short Form 10a | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  4-item measure of current physical function (range 1 to 5; higher scores = poorer physical function)
Patient-Reported Outcome Measurement Information System (PROMIS) - Emotional Distress - Anxiety - Short Form | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  4-item measure of anxiety symptoms in the past week (range 1 to 5; higher scores = more anxiety symptoms)
Patient-Reported Outcome Measurement Information System (PROMIS) - Emotional Distress - Depression - Short Form | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  4-item measure of depression symptoms in the past week (range 1 to 5; higher scores = more depression symptoms)
Patient Health Questionnaire - Depression | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  8-item measure of depression symptoms in the past week (range 0 to 3; higher scores = more depression symptoms)
Patient-Reported Outcome Measurement Information System (PROMIS) - Fatigue - Short Form | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  4-item measure of fatigue in the past week (range 1 to 5; higher scores = more fatigue)
Patient-Reported Outcome Measurement Information System (PROMIS) - Sleep Disturbance - Short Form | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  4-item measure of sleep disturbance in the past week (range 1 to 5; higher scores = more sleep disturbance)
Patient-Reported Outcome Measurement Information System (PROMIS) - Emotional Distress - Anger - Short Form 5a | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  5-item measure of anger in the past week (range 1 to 5; higher scores = more anger)
Positive and Negative Affect Schedule (PANAS) - Positive Affect - Short Form | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  5-item measure of positive affect in the past week (range 1 to 5; higher scores = more positive affectivity)
Posttraumatic Stress Disorder Checklist (PCL) - Short Form | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  5-item measure of trauma symptoms in the past week (range 1 to 4; higher scores = worse PTSD symptoms)
Pain Stages of Change Questionnaire (PSOCQ): Preparation and action | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  13-item measure on current readiness to adopt self-management for pain, Preparation and Action items only (range 1 to 5; higher scores = more ready to change)
Opioid Use | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  1-item measure on opioid use in past 7 days (range 1 to 7; higher scores = more days)
Employment | Baseline to post-treatment and 6-month follow-up
  3-item measure on current employment (options for current status and qualitative responses)
Post-Treatment Satisfaction Questionnaire | Post-Treatment to 6-Month Follow-Up
  8-item measure on patient post-treatment satisfaction (range 1 to 10; higher scores = more satisfied - also included qualitative responses)
Levels of Emotional Awareness Scale (LEAS) - Forms A and B | Baseline
  10-item measure of current emotional awareness (includes qualitative responses); responses coded for levels of emotional awareness; higher = greater awareness; Form A baseline and Form B at post-treatment
Other Pain Treatments and Health Care Use | Baseline to post-treatment and 6-month follow-up
  2-item measure of health care currently, the past 6 months, and the past 4 weeks (2 items with yes/no responses and remaining range 0 to 4; higher scores = more treatment)
Inventory of Interpersonal Problems (IIP) | Baseline to post-treatment and 6-month follow-up
  32-item measure of current interpersonal problems (range 0 to 4; higher scores = more interpersonal problems)
American College of Rheumatology (ACR) Fibromyalgia Diagnostic Criteria - 2011 | Baseline to post-treatment and 6-month follow-up
  8-item measure on fibromyalgia symptoms in the past week (items with yes/no responses, a checklist, and remaining range 0 to 3; higher scores = worse fibromyalgia symptoms)
Psychological Flexibility Scale (PSYFlex) | Baseline to post-treatment and 6-month follow-up
  6-item measure of psychological flexibility in the past week (range 0 to 5; higher scores = higher psychological flexibility)
The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool - Part II | Baseline to post-treatment and 6-month follow-up
  9-item measure on substance use in the past week (yes/no responses); higher scores = more use
Posttraumatic Stress Disorder Checklist (PCL) | Baseline to post-treatment and 6-month follow-up
  20-item measure of PTSD symptoms in the past month (range 0 to 4; higher scores = worse PTSD symptoms)

OTHER OUTCOMES:
Pain Catastrophizing Scale (PCS)-short form | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  Potential Mediator; 6-item measure of pain catastrophizing (range 0 to 4; higher scores = higher pain catastrophizing)
Pain Self-Efficacy Questionnaire (PSEQ) - Short Form | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  Potential Mediator; 4-item measure of current pain self-efficacy (range 0 to 6; higher scores = higher pain self-efficacy)
Survey of Pain Attitudes (SOPA): Pain Control, Disability, Harm, Emotion subscales | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  Potential Mediator; 4, 2-item measures of current pain attitudes (range 0 to 4; higher scores = more of that construct)
Behavioral Activation for Depression (BADS) - Short Form | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  Potential Mediator; 9-item measure of behavioral activation for depression in the past week (range 0 to 6; higher scores = higher behavioral activation)
Self-Compassion Scale (SCS) - Short Form | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  Potential Mediator; 12-item measure of situational self-compassion (range 1 to 5; higher scores = less self-compassion)
Chronic Pain Acceptance Questionnaire (CPAQ) | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  Potential Mediator; 8-item measure of current chronic pain acceptance (range 0 to 6; higher scores = more chronic pain acceptance)
Chronic Pain Values Inventory (CPVI) | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  Potential Mediator; 6-item measure of current values (checklist responses)
Emotional Approach Coping Scale (EAC) - Short Form | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  Potential Mediator; 4-item measure of emotional approach coping (range 1 to 4; higher scores = higher emotional approach coping)
Emotional Breakthrough Inventory (EBI) | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  Potential Mediator; 6-item measure of emotional breakthroughs in the past week (range 0 to 6; higher scores = more emotional breakthroughs)
Psychological Insight Questionnaire (PIQ) | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  Potential Mediator; 6-item measure of psychological insight in the past week (range 0 to 5; higher scores = more psychological insight)
Brain and Psychological Attributions for Pain | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  Potential Mediator; 9-item measure of current belief of brain and psychological attributions for pain (range 0 to 4; higher scores = higher belief in brain and psychological attributions for pain)
Pain Anxiety Symptom Scale (PASS) | Baseline to post-treatment and 6-month follow-up, and weekly during treatment
  Potential Mediator; 4-item measure of current pain anxiety symptoms (range 0 to 5; higher scores = worse pain anxiety symptoms)
Adverse Events | Weekly during treatment to post-treatment and 6-month follow-up
  Potential Mediator; 2-item measure of adverse events in the past week and past 6 months (checklist responses)
Working Alliance Inventory (WAI) - Patient | Weekly during treatment to post-treatment for three treatment arms only
  Potential Mediator; 6-item measure of current working alliance (range 0 to 5; higher scores = better working alliance)
Working Alliance Inventory (WAI) - Therapist - Short Form | Weekly during treatment to post-treatment for three treatment arms only
  Potential Mediator; 6-item measure of current working alliance (range 0 to 5; higher scores = better working alliance)
Therapist Checklist of Patient Engagement and Homework | Weekly during treatment to post-treatment for three treatment arms only
  Potential Mediator; 4-item measure on current patient engagement (range 0 to 8; higher scores = more patient engagement)
Treatment Expectancy and Credibility Questionnaire | Weekly during treatment to post-treatment for three treatment arms only
  Potential Mediator; 8-item measure on current treatment expectancy and credibility (range 0 to 10; higher scores = better treatment expectancy)

CONTACTS AND LOCATIONS:
Overall Officials: John W Burns, PhD, Principal Investigator — Rush University Medical Center
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Wayne State University, Detroit, Michigan

DOCUMENTS (2):
  • Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT06044649/SAP_000.pdf
  • Informed Consent Form (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/49/NCT06044649/ICF_001.pdf